CLINICAL TRIAL: NCT01892475
Title: TAKing Steps for Incentives (TAKSI) - A Randomized Controlled Trial to Motivate and Sustain Physical Activity Using Financial Incentives
Brief Title: TAKing Steps for Incentives
Acronym: TAKSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DPRT/AGE/2010/20
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Physical Activity; Incentives
Keywords: Physical Activity; Incentives; Mental Accounting; Older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cash Only (CO) (Experimental): As part of the Incentive-based physical activity program, drivers assigned to the Cash Only (CO) arm will earn incentives in the form of cash for meeting specified monthly step goals from Months 1 to 4.
  Interventions: Behavioral: Incentive-based physical activity program; Behavioral: 3-month follow up
- Mental-Accounting (MA) based (Experimental): As part of the Incentive-based physical activity program, drivers assigned to the Mental-Accounting (MA) based arm will receive incentives in the form of taxi rental credits for meeting specified monthly step goals from Months 1 to 4.
  Interventions: Behavioral: Incentive-based physical activity program; Behavioral: 3-month follow up

INTERVENTIONS:
Behavioral: Incentive-based physical activity program — Drivers will be offered rewards valued at a day's rental for meeting daily step targets over the specified number of days each month from Months 1 to 4, where steps will be tracked by a step counter. They will also be offered incentives for meeting the following criteria:
  1. Accurately predicting step target attainment the following months (SGD10)
  2. Wearing and providing step data over the month (SGD10 and a chance to win 1 of 3 cash prizes valued at SGD500)
Behavioral: 3-month follow up — After the 4-month RCT, drivers will be incentivized to wear the step counter for another 3 months (i.e. Months 5 to 7) to test if effects of the rewards are sustained once the reward is no longer in place. For wearing their step counter and providing their step data, drivers will receive a modest cash incentive (amounting to SGD10) each month as well as the chance to win 1 of 3 cash prizes valued at SGD500.

SUMMARY:
The purpose of this study is to test the overall effects of incentives on physical activity among older taxi drivers, and whether mental accounting exists in this context.

DETAILED DESCRIPTION:
As part of the 4-month Randomized Controlled Trial, participating taxi drivers will be assigned to 1 of 2 groups where they will receive either cash or taxi rental credits for meeting specified monthly step goals measured via a step counter. Subsequently, for an additional 3 months, drivers will be incentivized to wear step counters to test if effects of the rewards are sustained once the reward is no longer in place. Effects will be quantified in terms of step activity; and in terms of changes in Body Mass Index (BMI), Resting Heart Rate (HR), Blood Pressure (BP), self-reported General Health, Health-Related Quality of Life (HR-QOL) and work productivity.

ELIGIBILITY:
Inclusion Criteria:

* Must be a taxi driver who is a hirer, and who drives for at least 8 hours daily over 5 days
* Aged between 50 to 75
* English/Mandarin-speaking

Exclusion Criteria:

* Report difficulty doing 10 minutes of aerobic activities without stopping, walking up 10 stairs without stopping or performing basic activities of daily living
* Have any medical conditions that limit their ability to walk as a means of physical activity

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Steps taken | 7 months
  Steps will be assessed using Fitbit, which has an in-built 3-axis accelerometer that measures motion patterns. This will be evaluated monthly, from pre-Baseline through Month 7.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 7 months
  BMI will be evaluated using measured height and weight, and will be assessed at Months 0 (Baseline), 4 and 7.
Resting Heart Rate | 7 months
  Resting Heart Rate will be evaluated using a clinically validated machine (Welch Allyn SPOT Vital Signs Monitor), and will be assessed at Months 0 (Baseline), 4 and 7.
Blood Pressure | 7 months
  Blood pressure will be evaluated using a clinically validated machine (Welch Allyn SPOT Vital Signs Monitor), and will be assessed at Months 0 (Baseline), 4 and 7.
Self-reported General Health | 7 months
  Self-reported General Health will be evaluated using a validated survey instrument (SF12), and will be assessed at Months 0 (Baseline), 4 and 7.
Health-Related Quality of Life (HR-QOL) | 7 months
  Health-Related Quality of Life will be evaluated using a validated instrument (EQ-5D), and will be assessed at Months 0 (Baseline), 4 and 7.
Work Productivity | 7 months
  Work Productivity will be evaluated using a validated instrument (Work Productivity Activity Impairment Questionnaire) and other work-related data, and will be assessed throughout Months 0 (Baseline), 4 and 7.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Finkelstein, Ph.D, M.H.A., Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Graduate Medical School, Singapore, Singapore, Singapore